CLINICAL TRIAL: NCT01465464
Title: A Randomized, Double-Blind, Placebo-Controlled Phase III Trial Of TSU-68 In Combination With Transcatheter Arterial Chemoembolization In Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Orantinib In Combination With Transcatheter Arterial Chemoembolization In Patients With Unresectable Hepatocellular Carcinoma
Acronym: ORIENTAL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Taiho132150
Record Dates: First submitted 2011-11-01; First posted 2011-11-04 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — orantinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Orantinib (Experimental)
  Interventions: Drug: Orantinib (TSU-68)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orantinib (TSU-68) — 200 mg (1 tablet) of Orantinib was administered orally twice per day after meals, morning and evening.
  Arms: Orantinib
Drug: Placebo — 1 tablet was administered orally twice per day after meals, morning and evening.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the overall survival (OS) for Orantinib in combination with transcatheter arterial chemoembolization (TACE) versus placebo in combination with TACE in patients with unresectable hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
This is a randomized, multi-center, double-blind, placebo-controlled phase III trial of Orantinib administered in combination with TACE in patients with unresectable HCC.

Patients will be randomly assigned (1:1) to receive TACE given in combination with either Orantinib (200 mg orally, twice per day) or placebo.

ORIENTAL:ORantinib InvEstigatioN on TAce combination triaL.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed as HCC.
* Patients has no indications for treatment with curative hepatic resection or curative percutaneous local therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Patients are able to receive oral medication.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 888 (Actual)
Dates: Start 2010-12; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Pharmaceutical Co., Ltd., Study Director — Taiho Pharmaceutical Co., Ltd.
Locations (6):
- Japan (3):
  - Local Institution, Ōsaka-sayama, Osaka
  - Local Institution, Chuo-ku, Tokyo
  - Local Institution, Chiba
- South Korea (2):
  - Local Institution, Goyang-si, Gyeonggi-do
  - Local Institution, Seoul
- Local Institution, Taipei, Taiwan

REFERENCES:
- [Derived] Kudo M, Cheng AL, Park JW, Park JH, Liang PC, Hidaka H, Izumi N, Heo J, Lee YJ, Sheen IS, Chiu CF, Arioka H, Morita S, Arai Y. Orantinib versus placebo combined with transcatheter arterial chemoembolisation in patients with unresectable hepatocellular carcinoma (ORIENTAL): a randomised, double-blind, placebo-controlled, multicentre, phase 3 study. Lancet Gastroenterol Hepatol. 2018 Jan;3(1):37-46. doi: 10.1016/S2468-1253(17)30290-X. Epub 2017 Oct 4. PMID 28988687

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Orantinib | Placebo
Started | 444 | 444
Completed | 0 | 0
Not Completed | 444 | 444
Not completed — Adverse Event | 96 | 49
Not completed — Lack of Efficacy | 139 | 190
Not completed — Physician Decision | 13 | 5
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 46 | 30
Not completed — Other | 9 | 3
Not completed — Ongoing treatment at cutoff date | 140 | 166

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Orantinib | Placebo | Total
Number analyzed (Participants) | 444 | 444 | 888
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 189 | 202 | 391
  >=65 years | 255 | 242 | 497
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 80 | 161
  Male | 363 | 364 | 727
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 444 | 444 | 888
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 170 | 170 | 340
  Japan | 219 | 213 | 432
  Taiwan | 55 | 61 | 116

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival(OS)
Time Frame: The time from the date of enrollment to the date of death from any cause, assessed up to three years after randomizationof the last patient
Population: When approximately 50% of the targeted number of time to TACE discontinuation events were confirmed, interim analysis was performed by IDMC.
  Because the Committee considered that significant results would no longer be obtained, the IDMC recommended to the Sponsor that the clinical trial would be discontinued, and the Sponsor stopped this trial.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Orantinib | Placebo
Number analyzed (Participants) | 168 | 163
days | 946.0 [807.0 to 1050.0] | 984.0 [864.0 to NA] — The upper limit of median OS didn't reach.
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.435, Log Rank; Hazard Ratio (HR) = 1.090, 95% CI 2-sided [0.878 to 1.352]

2. Secondary Outcome: Time to Transcatheter Arterial Chemoembolization (TACE) Failure
Description: Patients should not receive additional TACE therapy in this study after meeting any of the following conditions, at the Investigator's discretion.
  1. The patient develops an intra-hepatic lesion that is uncontrolled by serial TACE
  2. Deterioration in arterial pathways to treat HCC that makes additional TACE impossible
  3. Severe vascular invasion occurs that makes additional TACE impossible
  4. Extra hepatic spread considered relevant to life expectancy that requires another treatment modality for HCC
  5. Liver function at grade Child-Pugh class C lasting for 28 days
Time Frame: The time from the date of enrollment to the date of event for TACE discontinuation, assessed up to three years after randomizationof the last patient
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Orantinib | Placebo
Number analyzed (Participants) | 174 | 206
days | 728.0 [604.0 to 813.0] | 602.0 [539.0 to 724.0]

ADVERSE EVENTS:
Time Frame: From the date of the first treatment to 30 days after the last treatment
Description: Main treatment discontinuation criteria
  * The Investigator concludes that the patients should be treated with another treatment modality except TACE for HCC
  * Patient has unacceptable/intolerable toxicities
  * Patient can not take both enhanced CT and enhanced MRI of the abdomen any more
  * Patient wishes to discontinue the treatment
Arm/Group | Orantinib | Placebo
All-Cause Mortality (participants affected / at risk) | 33/444 | 24/444
Serious Adverse Events (participants affected / at risk) | 200/444 | 134/444
Other Adverse Events (participants affected / at risk) | 443/444 | 436/444
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Orantinib (N=444) | Placebo (N=444)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Acute pericarditis (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0
Cardiopulmonary arrest (Cardiac disorders) | 1 | 0
Heart failure (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 3 | 0
Paroxysmal supraventricular tachycardia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Hydrocele cord (Congenital, familial and genetic disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 4 | 3
Cataract aggravated (Eye disorders) | 3 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1
Retinal macroaneurysm (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 9 | 7
Acute pancreatitis (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Acute gastric ulcer with haemorrhage (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 19 | 11
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 2
Duodenal ulcer (Gastrointestinal disorders) | 2 | 0
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 1 | 1
Epigastric pain (Gastrointestinal disorders) | 1 | 0
Esophageal hemorrhage (Gastrointestinal disorders) | 1 | 0
Esophageal varices hemorrhage (Gastrointestinal disorders) | 6 | 7
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric varices bleeding (Gastrointestinal disorders) | 1 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 2 | 7
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 1
Gastroesophageal varices hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 2
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 2
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Ischemia bowel (Gastrointestinal disorders) | 1 | 0
Ischemic enterocolitis (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Hematemesis (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 6 | 7
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Right upper quadrant pain (Gastrointestinal disorders) | 1 | 1
Ulcer duodenal haemorrhage (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1
Varices oesophageal (Gastrointestinal disorders) | 1 | 6
Vomiting (Gastrointestinal disorders) | 3 | 0
Condition aggravated (General disorders) | 1 | 0
Disease progression (General disorders) | 2 | 0
Edema limbs (General disorders) | 2 | 1
Fever (General disorders) | 13 | 11
Gait disturbance (General disorders) | 1 | 0
Malaise (General disorders) | 3 | 0
Multi organ failure (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Weakness generalised (General disorders) | 5 | 0
Fatigue (General disorders) | 0 | 2
Acute cholecystitis (Hepatobiliary disorders) | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 2 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 5
Biliary fistula (Hepatobiliary disorders) | 1 | 0
Biloma (Hepatobiliary disorders) | 5 | 1
Cholangitis (Hepatobiliary disorders) | 5 | 2
Cholangitis acute (Hepatobiliary disorders) | 1 | 2
Cholecystitis (Hepatobiliary disorders) | 3 | 4
Dilatation intrahepatic duct acquired (Hepatobiliary disorders) | 1 | 0
Gallbladder perforation (Hepatobiliary disorders) | 0 | 1
Haemobilia (Hepatobiliary disorders) | 0 | 2
Hepatic failure (Hepatobiliary disorders) | 16 | 11
Hepatic function disorder (Hepatobiliary disorders) | 11 | 4
Hepatic necrosis (Hepatobiliary disorders) | 1 | 1
Hepatopathy (Hepatobiliary disorders) | 0 | 2
Hyperbilirubinemia (Hepatobiliary disorders) | 1 | 2
Jaundice (Hepatobiliary disorders) | 1 | 2
Obstructive jaundice (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 2 | 2
Hepatic vein thrombosis (Hepatobiliary disorders) | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 6 | 0
Contrast media allergy (Immune system disorders) | 1 | 0
Acute bronchitis (Infections and infestations) | 1 | 0
Acute gastroenteritis (Infections and infestations) | 2 | 0
Acute pyelonephritis (Infections and infestations) | 2 | 0
Appendicitis perforated (Hepatobiliary disorders) | 2 | 1
Bacteremia (Hepatobiliary disorders) | 3 | 3
Biliary tract infection (Infections and infestations) | 1 | 3
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis of foot (Infections and infestations) | 1 | 0
Cryptococcal pneumonitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 1 | 0
Hepatic infection bacterial (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 2
Infectious colitis (Infections and infestations) | 1 | 1
Intra-abdominal infection (Infections and infestations) | 3 | 0
Liver abscess (Infections and infestations) | 34 | 3
Otitis media chronic (Infections and infestations) | 1 | 0
Periodontal abscess (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 5 | 1
Pulpitis (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 6 | 4
Spontaneous bacterial peritonitis (Infections and infestations) | 5 | 0
Tuberculous pleurisy (Infections and infestations) | 1 | 1
UTI (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Pyelonephritis (Infections and infestations) | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Fracture of lateral malleolus, closed (Injury, poisoning and procedural complications) | 2 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 0
Nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Polytraumatism (Injury, poisoning and procedural complications) | 1 | 0
Post embolization syndrome (Injury, poisoning and procedural complications) | 1 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 3 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 2
Traffic accident (Injury, poisoning and procedural complications) | 0 | 1
ALT increased (Investigations) | 3 | 1
AST increased (Investigations) | 3 | 1
Blood bilirubin increased (Investigations) | 1 | 2
CRP increased (Investigations) | 2 | 0
Creatinine increased (Investigations) | 2 | 1
Elevated liver enzymes (Investigations) | 1 | 0
Liver biopsy (Investigations) | 1 | 0
Spleen scan abnormal (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
WBC decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus aggravated (Metabolism and nutrition disorders) | 1 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Gout aggravated (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Investigations) | 2 | 1
Inappetence (Metabolism and nutrition disorders) | 2 | 0
Inappetence (Metabolism and nutrition disorders) | 1 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Cervical disc herniation (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in thigh (Musculoskeletal and connective tissue disorders) | 1 | 0
Pseudogout (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3 | 1
Wrist pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Avascular necrosis femoral head (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 3
Brain metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer of descending colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Hemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma non-resectable (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Hepatoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 6
Lung metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Spinal metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumor necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tumor rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of the gastrooesophageal junction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Cecal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Inverting papilloma of the nasal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm of cheek mucosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 5 | 5
Hepatic encephalopathy (Nervous system disorders) | 12 | 6
Intracranial hemorrhage (Nervous system disorders) | 3 | 1
Numbness of lower extremities (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Orientation disturbed (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 3
Renal failure (Renal and urinary disorders) | 4 | 4
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Gastrooesophageal variceal haemorrhage prophylaxis (Surgical and medical procedures) | 3 | 0
Induced abortion (Surgical and medical procedures) | 1 | 0
Oesophageal variceal ligation (Surgical and medical procedures) | 3 | 5
Varicose vein ruptured (Vascular disorders) | 1 | 0
Abdominal aortic aneurysm (Vascular disorders) | 0 | 1
Arterial stenosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Obstructive arteriosclerosis of lower extremities (Vascular disorders) | 0 | 1
Vascular disorder (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Orantinib (N=444) | Placebo (N=444)
Anaemia (Blood and lymphatic system disorders) | 54 | 32
Abdominal distension (Gastrointestinal disorders) | 50 | 53
Abdominal pain (Gastrointestinal disorders) | 317 | 292
Abdominal pain upper (Gastrointestinal disorders) | 56 | 46
Ascites (Gastrointestinal disorders) | 140 | 73
Constipation (Gastrointestinal disorders) | 179 | 147
Diarrhoea (Gastrointestinal disorders) | 123 | 70
Dyspepsia (Gastrointestinal disorders) | 51 | 47
Gastritis (Gastrointestinal disorders) | 23 | 29
Gastrointestinal pain (Gastrointestinal disorders) | 22 | 14
Nausea (Gastrointestinal disorders) | 179 | 179
Vomiting (Gastrointestinal disorders) | 126 | 116
Chills (General disorders) | 34 | 23
Face oedema (General disorders) | 138 | 8
Fatigue (General disorders) | 101 | 92
Malaise (General disorders) | 101 | 86
Non-cardiac chest pain (General disorders) | 32 | 25
Oedema peripheral (General disorders) | 130 | 59
Pyrexia (General disorders) | 264 | 284
Hepatic failure (Hepatobiliary disorders) | 24 | 20
Liver abscess (Infections and infestations) | 30 | 3
Upper respiratory tract infection (Infections and infestations) | 86 | 85
ALT increased (Investigations) | 200 | 170
AST increased (Investigations) | 223 | 189
ALP increased (Investigations) | 64 | 22
Bilirubin increased (Investigations) | 77 | 75
CRP increased (Investigations) | 47 | 44
Lymphocyte count decreased (Investigations) | 40 | 45
Platelet count decreased (Investigations) | 53 | 48
Weight decreased (Investigations) | 31 | 20
Decreased appetite (Metabolism and nutrition disorders) | 209 | 149
Hyperkalaemia (Metabolism and nutrition disorders) | 23 | 14
Hypoalbuminaemia (Metabolism and nutrition disorders) | 98 | 85
Hypokalaemia (Metabolism and nutrition disorders) | 34 | 16
Hyponatraemia (Metabolism and nutrition disorders) | 31 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 90 | 94
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 38 | 36
Myalgia (Musculoskeletal and connective tissue disorders) | 32 | 22
Pain in extremity (Musculoskeletal and connective tissue disorders) | 40 | 30
Dizziness (Nervous system disorders) | 38 | 35
Headache (Nervous system disorders) | 74 | 62
Insomnia (Psychiatric disorders) | 79 | 68
Chromaturia (Renal and urinary disorders) | 103 | 18
Proteinuria (Renal and urinary disorders) | 47 | 17
Hypertension (Vascular disorders) | 59 | 57
Cough (Respiratory, thoracic and mediastinal disorders) | 69 | 68
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 | 30
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 36 | 16
Pruritus (Skin and subcutaneous tissue disorders) | 43 | 51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other